CLINICAL TRIAL: NCT04767867
Title: Pre-oxygenation With Facemask Oxygen vs High-flow Nasal Oxygen vs High-flow Nasal Oxygen Plus Mouthpiece Oxygen - a Randomised Controlled Trial
Brief Title: Pre-oxygenation With Facemask Oxygen vs High-flow Nasal Oxygen vs High-flow Nasal Oxygen Plus Mouthpiece Oxygen
Acronym: PREOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, +Michael Callaghan - principal investigator, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Preox-HFNO
Record Dates: First submitted 2021-01-31; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Apnea; Respiration; Arrest; Anesthesia
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facemask oxygen (FM) (Experimental): 100% oxygen administered via facemask through circle system with adjustable pressure-limiting valve at 0 cmH20. Participant instructed to 'breathe normally'
  Interventions: Other: Pre-oxygenation
- High-flow nasal oxygen (HFNO) (Active Comparator): 100% oxygen administered via high-flow nasal cannulae at 50 L/min. Participant instructed to 'keep the mouth closed and breathe normally'
  Interventions: Other: Pre-oxygenation
- High-flow nasal oxygen plus mouthpiece oxygen (HFNO+MP) (Active Comparator): 100% oxygen administered via high-flow nasal cannulae at 50 L/min. Additionally, 100% oxygen administered via mouthpice through circle system with adjustable pressure-limiting valve at 0 cmH20. Participant instructed to 'keep the mouth closed and breathe normally'.
  Interventions: Other: Pre-oxygenation

INTERVENTIONS:
Other: Pre-oxygenation — Induction of anaesthesia after 2mins 45 seconds of pre-oxygenation with 1-1.5mcg/kg remifentanil plus 2-3mg/kg propofol. Propofol (10mg/kg/hr) and remifentanil (0.15mcg/kg/min) infusions commenced until study conclusion.
  Positive pressure ventilation commenced at Sp02 92%. Failure to intubate the patient during the first minute of apnoea results in withdrawal from the study.
  Blood samples obtained from an arterial catheter immediately prior to commencing pre-oxygenation, after 90 and 180 seconds of pre-oxygenation, after one minute of apnoea, and every two minutes during the apnoeic period.

SUMMARY:
Pre-oxygenation increases oxygen reserves in the body to reduce the likelihood of oxygen desaturation on induction of general anaesthesia. Pre-oxygenation with facemask is the commonest method method of pre-oxygenation. High-flow nasal oxygen is a newer alternative. This study randomises participants to receive pre-oxygenation by one of three methods: facemask, high-flow nasal oxygen, high-flow nasal oxygen plus mouthpiece.

DETAILED DESCRIPTION:
The administration of supplemental oxygen prior to induction of anaesthesia is known as pre-oxygenation. Pre-oxygenation increases oxygen reserves in the body with the purpose of delaying the time until oxygen desaturation after breathing stops (apnoea) following the administration of an anaesthetic. In the last decade, clinicians have begun utilising high-flow nasal oxygen for pre-oxygenation. However, the rationale for this is based largely on its ability to achieve ongoing oxygenation after the onset of apnoea (apnoeic oxygenation). This study isolates oxygen administration with high-flow nasal oxygen to the period when the person is breathing, without ongoing oxygen administration during the apnoea period, to quantify its effects during the pre-oxygenation period only. A third group of participants breathes oxygen through a mouthpiece in addition to receiving oxygen via high-flow nasal cannulae. The effect of these pre-oxygenation methods will be measured by the time taken until oxygen saturation levels decline to the lower end of the normal range (92%), along with other parameters such as blood oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ASA 1 or 2
* Receiving a general anaesthetic for non-emergent surgery

Exclusion Criteria:

* ASA score ≥3
* BMI ≥ 30 kg/m2
* Nasal obstruction
* Baseline SpO2 ≤95% on room air
* Anticipated difficult airway management
* Requirement for awake intubation
* Pregnancy
* Positive PCR test for coronavirus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Time to oxygen desaturation | Immediately after the intervention
  The time period from the onset of apnoea (determined by visual inspection) until an oxygen saturation of 92% is measured by pulse oximetry.

SECONDARY OUTCOMES:
Arterial partial pressure of oxygen after pre-oxygenation. | At 3 minutes of pre-oxygenation
  As measured by blood gas analysis
Arterial partial pressure of carbon dioxide change during pre-oxygenation | At 0 and 3 minutes
  As measured by blood gas analysis
Change in arterial partial pressure of carbon dioxide during apnoea | At 0, 1, 2 minutes and each 2 minutes thereafter
  As measured by blood gas analysis
Change in acid-base status during apnoea | At 0, 1, 2 minutes and each 2 minutes thereafter
  As measured by blood gas analysis
Correlation between end-tidal carbon dioxide measurement and arterial partial pressure of carbon dioxide | Etco2 obtained at the time of resumption of ventilation. Paco2 obtained from the preceding blood gas measurement.
  The EtCO2 value used for comparison is the highest value recorded during the first five respiratory cycles by manual ventilation with the adjustable pressure-limiting valve set at 20cmH20.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Callaghan, MB BCh BAO, Principal Investigator — Consultant Anaesthesiologist
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The sharing of anonymised patient-specific data that underlie results in any publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Post publication of results for up to fifteen years
Access Criteria: Investigator will consider requests to share patient-specific anonymised data in electronic format for the purpose of meta-analysis

REFERENCES:
- [Derived] Lyons C, McElwain J, Coughlan MG, O'Gorman DA, Harte BH, Kinirons B, Laffey JG, Callaghan M. Pre-oxygenation with facemask oxygen vs high-flow nasal oxygen vs high-flow nasal oxygen plus mouthpiece: a randomised controlled trial. Anaesthesia. 2022 Jan;77(1):40-45. doi: 10.1111/anae.15556. Epub 2021 Aug 17. PMID 34402044